CLINICAL TRIAL: NCT06390137
Title: The Immunomodulatory Effects of Frequency Specific Microcurrent In Obese Osteoarthritic Adults
Brief Title: Anti-Inflammatory Effects Of Frequency Specific Microcurrent (FSM) In Osteoarthritic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Samuel Spaiser, Principal Investigator, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2024-213-NSU
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FSM Treatment Group (Experimental): Participants receiving the 40 hertz/97 hertz alternating sharp square wave 200 uamp microcurrent treatment (machine is turned on and placed in an opaque bag to cover the screen; the machine is silent and therefore will be indistinguishable form placebo)
  Interventions: Device: Frequency Specific Microcurrent
- Placebo Group (Sham) (Placebo Comparator): Participants receiving sham microcurrent treatment (machine is turned off and placed in an opaque bag to cover the screen)
  Interventions: Device: Sham microcurrent treatment

INTERVENTIONS:
Device: Frequency Specific Microcurrent — The participant will receive an FSM treatment of 40 Hz on channel A and 97 Hz on channel B at 200 uamp with alternating current with a sharp square wave slope for 60 minutes with body contact points using a single towel wrapped posteriorly around the back at the level of T10 and the yellow (right side) and black (left side) leads will be attached to a second towel and wrapped anteriorly just below the abdomen and iliac crest. The TENS unit will be wrapped in an opaque bag so that the device is indistinguishable from that of the sham treatment.
  Other Names: E275 Transcutaneous Electrical Nerve Stimulator
  Arms: FSM Treatment Group
Device: Sham microcurrent treatment — The participant will receive a sham FSM treatment with the machine off wrapped in an opaque bag for 60 minutes with body contact points using a single towel wrapped posteriorly around the back at the level of T10 and the yellow (right side) and black (left side) leads will be attached to a second towel and wrapped anteriorly just below the abdomen and iliac crest.
  Other Names: E275 Transcutaneous Electrical Nerve Stimulator (Machine Off)
  Arms: Placebo Group (Sham)

SUMMARY:
It is hypothesized that application of frequency specific microcurrent can decrease inflammation in osteoarthritis patients resulting in decreased pain and potentially decrease disease progression. Participants will received the microcurrent treatment for one hour and a total of five blood draws to measure inflammatory markers. Participants will also complete a pre and post treatment pain questionnaire.

DETAILED DESCRIPTION:
After consent, the participant's height and weight will be measured and body mass index calculated using the Athena Health Patient Portal. Next, the participant will complete a pain questionnaire to capture their baseline level of pain as well as a sign a declaration stating that they have drank a quart of water in the past four hours. Then, the patient will have an intravenous port established in an antecubital vein.

The procedure that are being done for research purposed include five intravenous port blood draws and treatment with frequency specific microcurrent.

The patient will have an intravenous port established in an antecubital vein. A baseline 10 mL blood sample will be taken.

Randomization scheme is as follows - after the block size was determined, all possible balanced combinations of assignment within the block were calculated. Blocks were then randomly chosen to determine the patients' assignment into the groups.

An unblinded research coordinator with no other participation in the study will apply the randomization scheme (example included as attachment) to patients to receive either the active microcurrent treatment or a sham treatment. The active treatment includes turning on a Precision Distributing CustomCARE preprogrammed to produce 40 Hz on channel A and 97 Hz on channel B with 200 µamp alternating current polarity with a sharp square wave slope and placing it in an opaque bag so neither the participant or the study investigators know whether the device is on or off. The sham treatment involves not turning the device on and placing it in the same bag.

The electrical pulses will be sent from the CustomCARE through four, six-foot leads (red, green, yellow, and black) with alligator clips attached to two wet towels dampened with tap water. The participant will be seated in a comfortable chair, and the leads with the wet towels will be placed against bare skin as follows: the red (right side) and green (left side) leads will be attached to a single towel wrapped posteriorly around the back at the level of T10 and the yellow (right side) and black (left side) leads will be attached to a second towel and wrapped anteriorly just below the abdomen and iliac crest.

The participant will be instructed to relax for the next 60 minutes. 10mL of blood will be drawn from the IV port and collected in vacutainer plasma tubes before treatment and at the following timepoints during treatment: 15 minutes, 30 minutes, 45 minutes, 60 minutes. After completion of the treatment, the participant will complete a post-treatment pain scale questionnaire (duration 1 minute). Total study time per participant is two hours.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 29.9
* 18 years of age or older
* active osteoarthritis diagnosis

Exclusion Criteria:

* smoker
* BMI < 30
* have taken immune-enhancing dietary supplements or medications for inflammation in the past 10 days
* have or are currently being treated for any physician-diagnosed immune-modulating disease or disorder other than inflammatory arthritis
* received chemotherapy within the past year
* have ever received an FSM treatment with the frequency pair 40 Hz/97 Hz

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 | Baseline, during the intervention (15 minutes, 30 minutes, 45 minutes), and immediately after the intervention
  Plasma concentration

SECONDARY OUTCOMES:
Tumor Necrosis Factor Alpha | Baseline, during the intervention (15 minutes, 30 minutes, 45 minutes), and immediately after the intervention
  Plasma concentration
General Pain | Baseline, and immediately after the intervention
  0 - 10 Pain Scale, 10 being the worst pain imaginable and 0 being no pain at all

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Spaiser, MS, Principal Investigator — Nova Southeastern University College of Osteopathic Medicine
Locations (1):
- Robinson Family Clinic, Lakeland, Florida, United States

IPD SHARING:
Plan to Share IPD: No